CLINICAL TRIAL: NCT00661388
Title: A Single Arm, Open Label Study to Assess the Efficacy, Safety and Tolerability of Once-monthly Administration of Subcutaneous C.E.R.A. for the Treatment of Chronic Renal Anaemia in Pre-dialysis Patients Not Currently Treated With ESA.
Brief Title: A Study of Monthly Subcutaneous Mircera for the Treatment of Chronic Renal Anemia in Predialysis Patients Not Treated With ESA.
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Hoffmann-La Roche (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: ML21524
Record Dates: First submitted 2008-04-16; First posted 2008-04-18 (Estimated); Results first posted 2016-07-22 (Estimated); Last update posted 2025-09-11 (Actual); Status verified 2016-07

CONDITIONS: Anemia
MeSH Terms: conditions — Anemia | interventions — continuous erythropoietin receptor activator

ARMS (1):
- Continuous erythropoietin receptor activator (C.E.R.A.) (Experimental): Eligible participants will be administered C.E.R.A subcutaneously, every 4 weeks for 44 weeks. The initial dose of C.E.R.A. will be 1.2 micrograms/kilogram. Subsequent doses will be adjusted to maintain the individual participant's hemoglobin within the target range of 10.0 and 12.0 grams/deciliter.
  Interventions: Drug: methoxy polyethylene glycol-epoetin beta [Mircera]

INTERVENTIONS:
Drug: methoxy polyethylene glycol-epoetin beta [Mircera] — sc every month (starting dose 1.2 micrograms/kg)

SUMMARY:
This single arm study will assess the efficacy and safety of subcutaneous methoxy polyethylene glycol-epoetin beta (Mircera) for the correction and maintenance of hemoglobin levels in predialysis patients with renal anemia who are not currently treated with erythropoietin stimulating agents (ESA). Eligible patients will receive monthly subcutaneous injections of Mircera at an initial recommended dose of 1.2 micrograms/kg. The anticipated time on study treatment is 3-12 months, and the target sample size is 100-500 individuals.

ELIGIBILITY:
Inclusion Criteria:

* adult patients, >=18 years of age;
* chronic renal anemia;
* predialysis stage;
* no ESA therapy during previous 3 months.

Exclusion Criteria:

* transfusion of red blood cells during previous 2 months;
* poorly controlled hypertension requiring hospitalization in previous 6 months;
* significant acute or chronic bleeding.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 75 (Actual)
Dates: Start 2008-08; Primary Completion 2010-12 (Actual); Study Completion 2010-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Trials, Study Director — Hoffmann-La Roche
Locations (6):
- Turkey (Türkiye) (6):
  - Ankara
  - Denizli
  - Edirne
  - Istanbul
  - Kahramanmaraş
  - Konya

RESULTS

PARTICIPANT FLOW:
Recruitment Details: A total of 75 participants were enrolled in this study conducted from 12 August 2008 to December 2010 at 9 centers in Turkey.
Groups:
- C.E.R.A: Eligible participants were administered continuous erythropoietin receptor activator (C.E.R.A) subcutaneously, every 4 weeks for 44 weeks. The initial dose of C.E.R.A. was 1.2 micrograms (mcg)/kilogram (kg). Subsequent doses were adjusted to maintain the individual participant's hemoglobin (Hb) within the target range of 10.0 and 12.0 grams (g)/ deciliter (dL).
Period: Overall Study
Arm/Group | C.E.R.A
Started | 75
Completed | 51
Not Completed | 24
Not completed — Adverse Event | 14
Not completed — Protocol Violation | 7
Not completed — Renal transplantation | 1
Not completed — Dialysis initiation | 1
Not completed — Administrative reasons | 1

BASELINE CHARACTERISTICS:
Population: Safety population included all participants who received at least one dose of the trial medication and underwent a safety follow-up, whether withdrawn prematurely or not.
Groups:
- C.E.R.A: Eligible participants were administered C.E.R.A subcutaneously, every 4 weeks for 44 weeks. The initial dose of C.E.R.A. was 1.2 mcg/kg. Subsequent doses were adjusted to maintain the individual participant's Hb within the target range of 10.0 and 12.0 g/dL.
Arm/Group | C.E.R.A
Number analyzed (Participants) | 75
Age, Continuous [Mean (Standard Deviation); unit: years] | 52.8 (16.36)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 57
  Male | 18

OUTCOME MEASURES:

1. Primary Outcome: Mean Change in Hb Concentration Between Baseline and the Efficacy Evaluation Period
Description: Mean change in Hb concentration was calculated as the difference between the time adjusted average of Hb during the efficacy evaluation period (EEP [Week 29 to Week 36]), and the Hb at Baseline (Week 0). A positive change from baseline indicates improvement.
Time Frame: From Baseline (Week 0) to EEP (Week 29 to Week 36)
Population: Per protocol (PP) population included all participants who received at least one dose of C.E.R.A. and had at least one follow-up. Participants with less than three recorded Hb values during EEP; missing administration of C.E.R.A. during weeks 28-36; having inadequate iron status, were excluded.
Measure: Mean (Standard Deviation); unit: g/dL
Arm/Group | C.E.R.A
Number analyzed (Participants) | 41
g/dL | 1.99 (0.74)

2. Secondary Outcome: Mean Time to Achievement of Response During the EEP
Description: Participants with Hb concentrations within target range of 10-12 g/dl were considered to be responders. Mean time to achievement of response during the EEP (Week 29 to Week 36) is presented.
Time Frame: From Week 29 to Week 36
Population: PP population included all participants who received at least one dose of C.E.R.A. and had at least one follow-up. Participants with less than three recorded Hb values during EEP; missing administration of C.E.R.A. during weeks 28-36; having inadequate iron status, were excluded.
Measure: Mean (Standard Deviation); unit: Days
Arm/Group | C.E.R.A
Number analyzed (Participants) | 41
Days | 24.2 (20.96)

3. Secondary Outcome: The Percentage of Participants Whose Hb Concentrations Remained Within the Target Range of 10.0- 12.0 g/dLThroughout the EEP
Description: The percentage of participants whose Hb Concentrations remained within the target range of 10.0- 12.0 g/dL throughout the EEP (Week 29 to Week 36) is presented.
Time Frame: From Week 29 to Week 36
Population: PP population included all participants who received at least one dose of C.E.R.A. and had at least one follow-up variable were included. Participants with less than three recorded Hb values during EEP; participants missing administration of C.E.R.A. during weeks 28-36; participants with inadequate iron status, were excluded.
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | C.E.R.A
Number analyzed (Participants) | 41
Percentage of participants | 43.9 [28.5 to 60.3]

4. Secondary Outcome: Mean Time Spent by Participants in the Target Range of 10.0- 12.0 g/dL During the EEP
Description: Mean time spent by participants in the target range of 10.0- 12.0 g/dL during the EEP (Week 29 to Week 36) is presented.
Time Frame: From Week 29 to Week 36
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: Days
Arm/Group | C.E.R.A
Number analyzed (Participants) | 41
Days | 40.6 (16.31)

5. Secondary Outcome: Percentage of Participants Requiring Dose Adjustments During Dose Titration Period and EEP
Description: Percentage of participants requiring dose adjustments during dose titration period (DTP [Week 0 to Week 28]) and EEP (Week 29 to Week 36) is presented. The dose adjustments (increase or decrease) were required: if a single Hb concentration was either ≥ 13 g/dL or < 9 g/dL; if the difference of 2 consecutive Hb concentrations was ≥2 g/dL; if the values of scheduled Hb assessments on the day of administration of C.E.R.A. and on the previous study visit were both out of range of 10 to 12 g/dL; if the values of the scheduled Hb assessments on the day of administration of C.E.R.A. and on the previous study visit were both out of the range 10.5 to 11.5 g/dL. Dose adjustment could be made at any time at the discretion of the clinician if clinically warranted.
Time Frame: Weeks 0 to Week 36
Population: as for outcome 2
Measure: Number; unit: Percentage of participants
Arm/Group | C.E.R.A
Number analyzed (Participants) | 41
Percentage of participants
  Any dose adjustment in DTP | 85.4
  Dose increased in DTP | 14.6
  Dose decreased in DTP | 24.4
  Dose increased and decreased in DTP | 46.3
  Any dose adjustment in EEP | 56.1
  Dose increased in EEP | 17.1
  Dose decreased in EEP | 31.7
  Dose increased and decreased in EEP | 7.3

6. Secondary Outcome: Number of Participants Who Received Red Blood Cell Transfusions During the Study Period
Description: Red blood cell transfusions were given during the treatment period in case of medical need. Blood transfusions occurred during the DTP (Week 0 to Week 28), EEP (Week 29 to Week 36), and during the long term safety period (LSTP [Week 37 to Week 52]) are presented.
Time Frame: Up to Week 52
Population: Safety population included all participants who received at least one dose of the trial medication and underwent a safety follow-up, whether withdrawn prematurely or not. Number of participants who entered a particular phase is determined by 'n'.
Measure: Number; unit: Number of participants
Arm/Group | C.E.R.A
Number analyzed (Participants) | 75
Number of participants
  DTP (n = 75) | 2
  EEP (n = 57): number analyzed (Participants) | 57
  EEP (n = 57) | 1
  LSTP (n = 54): number analyzed (Participants) | 54
  LSTP (n = 54) | 1

7. Secondary Outcome: Number of Participants Who Experienced Any Adverse Events or Serious Adverse Events
Description: An adverse event (AE) is any untoward medical occurrence in a participant or clinical investigation participant administered a pharmaceutical product and which does not necessarily have to have a causal relationship with this treatment. An AE can therefore be any unfavorable and unintended sign (including an abnormal laboratory finding), symptom, or disease temporally associated with the use of a medicinal product, whether or not considered related to the medicinal product. A serious adverse event (SAE) is any untoward medical occurrence that at any dose results in death, are life threatening, requires hospitalization or prolongation of hospitalization or results in disability/incapacity, and congenital anomaly/birth defect.
Time Frame: Up to Week 52
Population: as for baseline characteristics
Measure: Number; unit: Participants
Arm/Group | C.E.R.A
Number analyzed (Participants) | 75
Participants
  Any AEs | 58
  Any SAEs | 24

8. Secondary Outcome: Mean Change From Baseline in Hb Concentration Over Time
Description: Mean change from Baseline in Hb concentration was calculated as the difference between Baseline and post-baseline measurements. It was recorded for each participant at enrollment (Week 0) and at different time points during the study up to Week 48.
Time Frame: Baseline (Week 0), Weeks 8, 16, 24, 32, 40, and 48
Population: Safety population included all participants who received at least one dose of the trial medication and underwent a safety follow-up, whether withdrawn prematurely or not. Number of participants analyzed at a particular visit is determined by 'n'.
Measure: Mean (Standard Deviation); unit: g/dL
Arm/Group | C.E.R.A
Number analyzed (Participants) | 70
g/dL
  Week 8 (n = 70) | 1.50 (0.96)
  Week 16 (n = 62): number analyzed (Participants) | 62
  Week 16 (n = 62) | 2.03 (1.16)
  Week 24 (n = 59): number analyzed (Participants) | 59
  Week 24 (n = 59) | 1.86 (1.01)
  Week 32 (n = 55): number analyzed (Participants) | 55
  Week 32 (n = 55) | 1.85 (0.84)
  Week 40 (n = 52): number analyzed (Participants) | 52
  Week 40 (n = 52) | 1.84 (1.06)
  Week 48 (n = 48): number analyzed (Participants) | 48
  Week 48 (n = 48) | 1.59 (0.81)

9. Secondary Outcome: Mean Change From Baseline in Hematocrit Level Over Time
Description: Mean change from Baseline in hematocrit level was calculated as the difference between Baseline and post-baseline measurements. It was recorded for each participant at enrollment (Week 0) and at different time points during the study up to Week 48.
Time Frame: Baseline (Week 0), Weeks 8, 16, 24, 32, 40, and 48
Population: as for outcome 8
Measure: Mean (Standard Deviation); unit: Fraction
Arm/Group | C.E.R.A
Number analyzed (Participants) | 70
Fraction
  Week 8 (n = 70) | 0.05 (0.03)
  Week 16 (n = 62): number analyzed (Participants) | 62
  Week 16 (n = 62) | 0.06 (0.04)
  Week 24 (n = 59): number analyzed (Participants) | 59
  Week 24 (n = 59) | 0.06 (0.03)
  Week 32 (n = 55): number analyzed (Participants) | 55
  Week 32 (n = 55) | 0.06 (0.03)
  Week 40 (n = 51): number analyzed (Participants) | 51
  Week 40 (n = 51) | 0.06 (0.03)
  Week 48 (n = 49): number analyzed (Participants) | 49
  Week 48 (n = 49) | 0.05 (0.02)

10. Secondary Outcome: Mean Change From Baseline in Erythrocyte Mean Corpuscular Volume Over Time
Description: Mean change from Baseline in erythrocyte mean corpuscular volume was calculated as the difference between Baseline and post-baseline measurements. It was recorded for each participant at enrollment (Week 0) and at different time points during the study up to Week 48.
Time Frame: Baseline (Week 0), Weeks 8, 16, 24, 32, and 48
Population: as for outcome 8
Measure: Mean (Standard Deviation); unit: Femtoliters
Arm/Group | C.E.R.A
Number analyzed (Participants) | 65
Femtoliters
  Week 8 (n = 65) | 0.17 (3.20)
  Week 16 (n = 57): number analyzed (Participants) | 57
  Week 16 (n = 57) | -1.31 (3.70)
  Week 24 (n = 55): number analyzed (Participants) | 55
  Week 24 (n = 55) | -1.10 (4.40)
  Week 32 (n = 52): number analyzed (Participants) | 52
  Week 32 (n = 52) | -0.34 (4.62)
  Week 48 (n = 47): number analyzed (Participants) | 47
  Week 48 (n = 47) | 0.97 (3.67)

11. Secondary Outcome: Mean Change From Baseline in White Blood Cells and Platelets Concentrations Over Time
Description: Mean change from Baseline in white blood cells (WBCs) and platelets concentrations was calculated as the difference between Baseline and post-baseline measurements. It was recorded for each participant at enrollment (Week 0) and at different time points during the study up to Week 48.
Time Frame: Baseline (Week 0), Weeks 8, 16, 24, 32, 40, and 48
Population: as for outcome 8
Measure: Mean (Standard Deviation); unit: 10^9 cells/Liter (L)
Arm/Group | C.E.R.A
Number analyzed (Participants) | 66
10^9 cells/Liter (L)
  WBCs at Week 8 (n = 66) | 0.04 (1.59)
  WBCs at Week 16 (n = 58): number analyzed (Participants) | 58
  WBCs at Week 16 (n = 58) | 0.06 (1.36)
  WBCs at Week 24 (n = 55): number analyzed (Participants) | 55
  WBCs at Week 24 (n = 55) | 0.12 (1.46)
  WBCs at Week 32 (n = 52): number analyzed (Participants) | 52
  WBCs at Week 32 (n = 52) | 0.01 (1.48)
  WBCs at Week 40 (n = 47): number analyzed (Participants) | 47
  WBCs at Week 40 (n = 47) | -0.13 (1.54)
  WBCs at Week 48 (n = 47): number analyzed (Participants) | 47
  WBCs at Week 48 (n = 47) | 0.04 (1.43)
  Platelets at Week 8 (n = 66) | -8.39 (52.64)
  Platelets at Week 16 (n = 58): number analyzed (Participants) | 58
  Platelets at Week 16 (n = 58) | -15.73 (46.37)
  Platelets at Week 24 (n = 55): number analyzed (Participants) | 55
  Platelets at Week 24 (n = 55) | -20.55 (41.59)
  Platelets at Week 32 (n = 52): number analyzed (Participants) | 52
  Platelets at Week 32 (n = 52) | -25.34 (47.22)
  Platelets at Week 40 (n = 47): number analyzed (Participants) | 47
  Platelets at Week 40 (n = 47) | -25.84 (46.90)
  Platelets at Week 48 (n = 47): number analyzed (Participants) | 47
  Platelets at Week 48 (n = 47) | -23.40 (40.74)

12. Secondary Outcome: Mean Change From Baseline in Albumin Concentration Over Time
Description: Mean change from Baseline in albumin concentration was calculated as the difference between Baseline and post-baseline measurements. It was recorded for each participant at enrollment (Week 0) and at different time points during the study up to Week 48.
Time Frame: Baseline (Week 0), Weeks 8, 16, 24, 32, 40, and 48
Population: as for outcome 8
Measure: Mean (Standard Deviation); unit: g/L
Arm/Group | C.E.R.A
Number analyzed (Participants) | 62
g/L
  Week 8 (n = 62) | 0.45 (3.12)
  Week 16 (n = 52): number analyzed (Participants) | 52
  Week 16 (n = 52) | 0.06 (3.27)
  Week 24 (n = 53): number analyzed (Participants) | 53
  Week 24 (n = 53) | -0.30 (3.59)
  Week 32 (n = 48): number analyzed (Participants) | 48
  Week 32 (n = 48) | 0.24 (5.37)
  Week 40 (n = 45): number analyzed (Participants) | 45
  Week 40 (n = 45) | -0.57 (3.34)
  Week 48 (n = 46): number analyzed (Participants) | 46
  Week 48 (n = 46) | -0.61 (3.82)

13. Secondary Outcome: Mean Change From Baseline in C-Reactive Protein Concentration Over Time
Description: Mean change from Baseline in C-Reactive Protein concentration was calculated as the difference between Baseline and post-baseline measurements. It was recorded for each participant at enrollment (Week 0) and at different time points during the study up to Week 48.
Time Frame: Baseline (Week 0), Weeks 8, 16, 24, 32, 40, and 48
Population: as for outcome 8
Measure: Mean (Standard Deviation); unit: Milligrams /L
Arm/Group | C.E.R.A
Number analyzed (Participants) | 55
Milligrams /L
  Week 8 (n = 55) | -1.82 (13.24)
  Week 16 (n = 44): number analyzed (Participants) | 44
  Week 16 (n = 44) | -1.80 (13.05)
  Week 24 (n = 45): number analyzed (Participants) | 45
  Week 24 (n = 45) | 0.03 (9.31)
  Week 32 (n = 38): number analyzed (Participants) | 38
  Week 32 (n = 38) | -0.33 (9.88)
  Week 40 (n = 42): number analyzed (Participants) | 42
  Week 40 (n = 42) | -1.49 (4.78)
  Week 48 (n = 39): number analyzed (Participants) | 39
  Week 48 (n = 39) | 0.86 (6.57)

14. Secondary Outcome: Mean Change From Baseline in Phosphate and Potassium Concentrations Over Time
Description: Mean change from Baseline in phosphate and potassium concentrations was calculated as the difference between Baseline and post-baseline measurements. It was recorded for each participant at enrollment (Week 0) and at different time points during the study up to Week 48.
Time Frame: Baseline (Week 0), Weeks 8, 16, 24, 32, 40, and 48
Population: as for outcome 8
Measure: Mean (Standard Deviation); unit: Millimoles /L
Arm/Group | C.E.R.A
Number analyzed (Participants) | 63
Millimoles /L
  Phosphate at Week 8 (n = 59): number analyzed (Participants) | 59
  Phosphate at Week 8 (n = 59) | 0.11 (0.35)
  Phosphate at Week 16 (n = 48): number analyzed (Participants) | 48
  Phosphate at Week 16 (n = 48) | 0.06 (0.26)
  Phosphate at Week 24 (n = 51): number analyzed (Participants) | 51
  Phosphate at Week 24 (n = 51) | 0.07 (0.36)
  Phosphate at Week 32 (n = 45): number analyzed (Participants) | 45
  Phosphate at Week 32 (n = 45) | 0.13 (0.27)
  Phosphate at Week 40 (n = 44): number analyzed (Participants) | 44
  Phosphate at Week 40 (n = 44) | 0.06 (0.31)
  Phosphate at Week 48 (n = 43): number analyzed (Participants) | 43
  Phosphate at Week 48 (n = 43) | 0.07 (0.30)
  Potassium at Week 8 (n = 63) | 0.12 (0.53)
  Potassium at Week 16 (n = 54): number analyzed (Participants) | 54
  Potassium at Week 16 (n = 54) | 0.03 (0.68)
  Potassium at Week 24 (n = 53): number analyzed (Participants) | 53
  Potassium at Week 24 (n = 53) | 0.02 (0.56)
  Potassium at Week 32 (n = 49): number analyzed (Participants) | 49
  Potassium at Week 32 (n = 49) | -0.04 (0.63)
  Potassium at Week 40 (n = 46): number analyzed (Participants) | 46
  Potassium at Week 40 (n = 46) | 0.16 (0.56)
  Potassium at Week 48 (n = 47): number analyzed (Participants) | 47
  Potassium at Week 48 (n = 47) | 0.03 (0.70)

15. Secondary Outcome: Mean Change From Baseline in Total Iron Binding Capacity and Iron Concentrations Over Time
Description: Mean change from Baseline in total iron binding capacity (TIBC) and iron concentrations was calculated as the difference between Baseline and post-baseline measurements. It was recorded for each participant at enrollment (Week 0) and at different time points during the study up to Week 48.
Time Frame: Baseline (Week 0), Weeks 8, 16, 24, 32, 40, and 48
Population: as for outcome 8
Measure: Mean (Standard Deviation); unit: Micromole /L
Arm/Group | C.E.R.A
Number analyzed (Participants) | 63
Micromole /L
  TIBC at Week 8 (n = 62): number analyzed (Participants) | 62
  TIBC at Week 8 (n = 62) | 0.09 (10.02)
  TIBC at Week 16 (n = 53): number analyzed (Participants) | 53
  TIBC at Week 16 (n = 53) | -0.21 (8.12)
  TIBC at Week 24 (n = 52): number analyzed (Participants) | 52
  TIBC at Week 24 (n = 52) | 0.34 (10.78)
  TIBC at Week 32 (n = 47): number analyzed (Participants) | 47
  TIBC at Week 32 (n = 47) | 0.15 (10.53)
  TIBC at Week 40 (n = 45): number analyzed (Participants) | 45
  TIBC at Week 40 (n = 45) | 2.24 (19.75)
  TIBC at Week 48 (n = 46): number analyzed (Participants) | 46
  TIBC at Week 48 (n = 46) | -2.02 (11.05)
  Iron at Week 8 (n = 63) | -1.93 (7.31)
  Iron at Week 16 (n = 53): number analyzed (Participants) | 53
  Iron at Week 16 (n = 53) | 0.31 (6.79)
  Iron at Week 24 (n = 54): number analyzed (Participants) | 54
  Iron at Week 24 (n = 54) | 0.55 (8.56)
  Iron at Week 32 (n = 47): number analyzed (Participants) | 47
  Iron at Week 32 (n = 47) | 0.68 (8.64)
  Iron at Week 40 (n = 45): number analyzed (Participants) | 45
  Iron at Week 40 (n = 45) | 1.64 (6.76)
  Iron at Week 48 (n = 46): number analyzed (Participants) | 46
  Iron at Week 48 (n = 46) | 0.80 (9.24)

16. Secondary Outcome: Mean Change From Baseline in Creatinine Concentration Over Time
Description: Mean change from Baseline in creatinine concentration was calculated as the difference between Baseline and post-baseline measurements. It was recorded for each participant at enrollment (Week 0) and at different time points during the study up to Week 48.
Time Frame: Baseline (Week 0), Weeks 8, 16, 32, 40
Population: as for outcome 8
Measure: Median (Full Range); unit: Micromole/L
Arm/Group | C.E.R.A
Number analyzed (Participants) | 4
Micromole/L
  Week 8 (n = 4) | 23.87 [-24.8 to 44.2]
  Week 16 (n = 2): number analyzed (Participants) | 2
  Week 16 (n = 2) | 123.67 [53.0 to 194.5]
  Week 32 (n = 2): number analyzed (Participants) | 2
  Week 32 (n = 2) | -8.40 [-17.7 to 0.9]
  Week 40 (n = 1): number analyzed (Participants) | 1
  Week 40 (n = 1) | 17.7 [17.7 to 17.7]

17. Secondary Outcome: Mean Change From Baseline in Ferritin Concentration Over Time
Description: Mean change from Baseline in ferritin concentration was calculated as the difference between Baseline and post-baseline measurements. It was recorded for each participant at enrollment (Week 0) and at different time points during the study up to Week 48.
Time Frame: Baseline (Week 0), Weeks 8, 16, 24, 32, 40, and 48
Population: as for outcome 8
Measure: Mean (Standard Deviation); unit: mcg/L
Arm/Group | C.E.R.A
Number analyzed (Participants) | 52
mcg/L
  Ferritin at Week 8 (n = 52) | -95.15 (86.09)
  Ferritin at Week 16 (n = 49): number analyzed (Participants) | 49
  Ferritin at Week 16 (n = 49) | -82.82 (115.68)
  Ferritin at Week 24 (n = 42): number analyzed (Participants) | 42
  Ferritin at Week 24 (n = 42) | -71.98 (131.47)
  Ferritin at Week 32 (n = 39): number analyzed (Participants) | 39
  Ferritin at Week 32 (n = 39) | -78.45 (121.12)
  Ferritin at Week 40 (n = 42): number analyzed (Participants) | 42
  Ferritin at Week 40 (n = 42) | -59.94 (141.89)
  Ferritin at Week 48 (n = 43): number analyzed (Participants) | 43
  Ferritin at Week 48 (n = 43) | -43.46 (146.58)

18. Secondary Outcome: Mean Change From Baseline in Transferrin Saturation Over Time
Description: Mean change from Baseline in transferrin saturation (TSAT) was calculated as the difference between Baseline and post-baseline measurements. It was recorded for each participant at enrollment (Week 0) and at different time points during the study up to Week 48.
Time Frame: Baseline (Week 0), Weeks 8, 16, 24, 32, 40, and 48
Population: as for outcome 8
Measure: Mean (Standard Deviation); unit: Percentage of Transferrin Saturation
Arm/Group | C.E.R.A
Number analyzed (Participants) | 62
Percentage of Transferrin Saturation
  TSAT at Week 8 (n = 62) | -5.91 (19.83)
  TSAT at Week 16 (n = 52): number analyzed (Participants) | 52
  TSAT at Week 16 (n = 52) | 1.69 (13.85)
  TSAT at Week 24 (n = 51): number analyzed (Participants) | 51
  TSAT at Week 24 (n = 51) | 1.42 (15.15)
  TSAT at Week 32 (n = 47): number analyzed (Participants) | 47
  TSAT at Week 32 (n = 47) | 2.52 (15.70)
  TSAT at Week 40 (n = 45): number analyzed (Participants) | 45
  TSAT at Week 40 (n = 45) | 3.52 (13.02)
  TSAT at Week 48 (n = 46): number analyzed (Participants) | 46
  TSAT at Week 48 (n = 46) | 5.32 (21.60)

ADVERSE EVENTS:
Time Frame: Up to Week 52
Description: SAEs and non-serious AEs were reported for the safety population, comprised of participants who received at least one dose of study drug, whether withdrawn prematurely or not, and who had at least one follow-up data point.
Arm/Group | C.E.R.A
Serious Adverse Events (participants affected / at risk) | 24/75
Other Adverse Events (participants affected / at risk) | 38/75
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | C.E.R.A (N=75)
Thrombocytosis (Blood and lymphatic system disorders) | 1
Angina pectoris (Cardiac disorders) | 2
Coronary artery disease (Cardiac disorders) | 1
Atrial septal defect (Congenital, familial and genetic disorders) | 1
Nausea (Gastrointestinal disorders) | 1
Chest pain (General disorders) | 1
Oedema (General disorders) | 1
Gastroenteritis (Infections and infestations) | 1
Pyelonephritis acute (Infections and infestations) | 1
Foot fracture (Injury, poisoning and procedural complications) | 1
Hip fracture (Injury, poisoning and procedural complications) | 1
Blood creatine increased (Investigations) | 2
Blood creatinine increased (Investigations) | 1
Creatinine renal clearance decreased (Investigations) | 1
Diabetic foot (Metabolism and nutrition disorders) | 1
Hypervolaemia (Metabolism and nutrition disorders) | 1
Metabolic acidosis (Metabolism and nutrition disorders) | 6
Azotaemia (Renal and urinary disorders) | 1
Renal failure (Renal and urinary disorders) | 1
Renal failure acute (Renal and urinary disorders) | 1
Dyspnoea exertional (Respiratory, thoracic and mediastinal disorders) | 1
Haemodialysis (Surgical and medical procedures) | 1
Insertion of ambulatory peritoneal catheter (Surgical and medical procedures) | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | C.E.R.A (N=75)
Hypertension (Vascular disorders) | 15
Constipation (Gastrointestinal disorders) | 7
Nausea (Gastrointestinal disorders) | 6
Hyperkalaemia (Metabolism and nutrition disorders) | 9
Hyperlipidaemia (Metabolism and nutrition disorders) | 4
Urinary tract infection (Infections and infestations) | 6
Hyperparathyroidism secondary (Endocrine disorders) | 5
Blood pressure increased (Investigations) | 4
Back pain (Musculoskeletal and connective tissue disorders) | 4

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The Study being conducted under this Agreement is part of the Overall Study. Investigator is free to publish in reputable journals or to present at professional conferences the results of the Study, but only after the first publication or presentation that involves the Overall Study. The Sponsor may request that Confidential Information be deleted and/or the publication be postponed in order to protect the Sponsor's intellectual property rights.